CLINICAL TRIAL: NCT01590134
Title: Pilot Studies on the Efficacy and Safety of Dietary Iron Supplementation
Brief Title: The Efficacy and Safety of Iron Supplementation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLS/2012/1
Record Dates: First submitted 2012-04-30; First posted 2012-05-02 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2012-04

CONDITIONS: Healthy
Keywords: volunteers; Pilot study; There are no pre registration evaluations.; Inclusion criteria: to be a healthy, consenting volunteer not currently receiving iron supplements.; Exclusion criteria: 1) Needle phobia; 2) Currently receiving iron supplements; 3) Unable to provide informed consent
MeSH Terms: interventions — ferrous sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Following randomisation,to no active intervention, blood and urine samples will be collected at 6 stated intervals over a 48 hour period
  Total number of participants in arm = 6
- Iron control (Active Comparator): Following randomisation, on each of two consecutive mornings, the participant will receive a single dose of ferrous sulphate 200mg. Blood and urine samples will be collected pre first dose, and at 5 further stated intervals over a 48 hour period.
  Total number of participants in arm = 6
  Interventions: Drug: Ferrous sulphate
- Dietary supplement (Experimental): Following randomisation, on each of two consecutive mornings, the participant will receive the experimental dietary iron supplement. Blood and urine samples will be collected pre first dose, and at 5 further stated intervals over a 48 hour period.
  Toal participants in arm = 6
  Interventions: Dietary Supplement: Dietary supplement of iron

INTERVENTIONS:
Dietary Supplement: Dietary supplement of iron — 1 tablespoon of a dietary iron supplement containing 2.64mg of elemental iron
  Arms: Dietary supplement
Drug: Ferrous sulphate — 200mg coated dried tablet containing 65mg elemental iron, equivalent to prophylactic daily dose as defined by the British National Formulary
  Arms: Iron control

SUMMARY:
Each year, 5 million packs of iron tablets are dispensed in England and Wales to treat anaemia due to iron deficiency. Iron tablets are not always easy to take. The investigators think that there could be ways to reduce the number of iron tablets needed, by increasing the dietary intake of iron. In this study the investigators will assess the efficacy and safety of a dietary iron supplement compared to iron tablets using controls and new biomarkers.

DETAILED DESCRIPTION:
18 healthy individuals will be randomised to one of three arms, and for two consecutive mornings, will receive either an iron tablet (ferrous sulphate 200mg), a dietary iron supplement, or no agent.

Blood and urine samples will be collected pre-dose, and at stated intervals 2.5, 4, 7, 24 and 48 hours post first dose.

The standard deviations of data obtained in this pilot study will be used to perform power calculations for our future studies in this field.

ELIGIBILITY:
Inclusion Criteria:

To be a healthy, consenting volunteer not currently receiving iron supplements.

Exclusion Criteria:

1. Needle phobia
2. Currently receiving iron supplements
3. Unable to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Iron levels in blood tests | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Claire L Shovlin, PhD MA MB BChir FRCP, Principal Investigator — Imperial College London
Locations (1):
- Wellcome Trust-McMichael Clinical Research Facility, Imperial college London, London, United Kingdom

REFERENCES:
- [Background] Further analyses are in progress for full manuscript.
- [Result] Gilson C, Busbridge M, Shovlin CL, Iron tablet profiling. Hematology Reports 2013: 5 (s1),30-1